CLINICAL TRIAL: NCT01633307
Title: Effect of a Nationwide Teaching Program on the Frequency of Inappropriate Intravenous Lines in Internal Medicine: A Randomized Controlled Trial
Brief Title: Decrease the Frequency of Inappropriate Intravenous Lines in Internal Medicine
Acronym: PERMI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hopital Lariboisière (Other)
Responsible Party: Principal Investigator, Stephane Mouly, MD PhD, Professor of Medicine, Hopital Lariboisière
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: PERMI
Record Dates: First submitted 2012-06-19; First posted 2012-07-04 (Estimated); Last update posted 2012-07-04 (Estimated); Status verified 2012-06

CONDITIONS: Acute Medical Patients Hospitalized in Internal Medicine
Keywords: education; intravenous infusion
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental (Experimental): Intervention (Teaching program)
  Interventions: Other: Education
- Control group (No Intervention): No teaching program

INTERVENTIONS:
Other: Education — Teaching program
  Arms: Experimental

SUMMARY:
Aim: to determine whether a nationwide teaching program delivered to medical doctors can decrease the use of inappropriate intravenous lines in internal medicine

DETAILED DESCRIPTION:
Nationwide multicentre randomized prospective controlled trial enrolling 59 french internal medicine departments. During the first study visit, we collected data of patients with intravenous infusions from each participating centre in order to determine the number and frequency of inappropriate intravenous lines. Using a computerized randomization process (on a 1:1 basis), the participating centres were randomized; Half centres (interventional group) received an educational program consisting of educational material and two educational sessions; the other half did not receive the educational program (control group). The educational program provided medical doctors with posters and slides containing information on valid indications for the prescription and use of intravenous infusions (inability to drink or eat, malabsorption, medication only available intravenously with no oral equivalent). Based on a previous pilot study, we assumed that the the frequency of inappropriate intravenous lines with be approximately 20% at baseline and hypothesize that the nationwide teaching program will decrease this frequency by 50%.

ELIGIBILITY:
Inclusion Criteria:

* Internal medicine department

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2007-01; Primary Completion 2007-04 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
frequency of inappropriate intravenous infusion in internal medicine department

CONTACTS AND LOCATIONS:
Overall Officials: stephane J mouly, MD PhD, Principal Investigator — Hopital Lariboisiere

REFERENCES:
- [Derived] Champion K, Mouly S, Lloret-Linares C, Lopes A, Vicaut E, Bergmann JF; PERMI Investigators Committee. Optimizing the use of intravenous therapy in internal medicine. Am J Med. 2013 Oct;126(10):925.e1-9. doi: 10.1016/j.amjmed.2013.03.028. Epub 2013 Aug 3. PMID 23920107